CLINICAL TRIAL: NCT06652893
Title: Real-world Efficacy and Safety of Sinovial®HL Single Injection in the Treatment of Symptomatic Knee Osteoarthritis: an Observational Study
Brief Title: Efficacy and Safety of Sinovial®HL Single Injection in the Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Marcin Domżalski (Other)
Collaborators: IBSA Institut Biochimique SA (Industry)
Responsible Party: Sponsor-Investigator, Marcin Domżalski, Principal Investigator, Sporto Clinic
Organization: Sporto Clinic (Other)
Other Study IDs: K.B. 22/2022
Record Dates: First submitted 2024-10-17; First posted 2024-10-22 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Osteoarthritis of Knee
Keywords: knee osteoarthritis; hialuronic acid; knee function
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Fifty consecutive patients who met the inclusion criteria participated in the study: Consecutive patients with knee osteoarthritis and with a medical indication for viscosupplementation with hybrid hialuronic acid (HA) who fulfilled the inclusion criteria were recruited for the study. The inclusion criteria were: a medical indication for viscosupplementation therapy with hybrid HA; patients aged between 45 and 80 years; diagnosis of femorotibial gonarthrosis associated with femoro-patellar arthrosis or isolated, gonarthrosis symptoms for at least 6 months; patients who failed to respond to analgesics and/or regular NSAIDs, or were proved to be intolerant to the regular use of analgesics, NSAIDS, or weak opioids; grade 2 to 3 OA in the Kellgren-Lawrence grading scale ; pain when walking measured by the Visual Analog Scale of at least 40 mm on the targeted knee; and contralateral knee pain when walking with aVAS of less than 10 mm. The exclusion criteria were: inability to understand the aim of the study, inability to provide acceptable consent, pregnancy, serious ps
  Interventions: Drug: Sinovial

INTERVENTIONS:
Drug: Sinovial — A single intra-articular injection of hybrid HA complex, Sinovial® HL (IBSA Pharmaceuticals, Italy, patent number WO/2012/032151 ) in the knee was performed from the lateral approach to the suprapatellar recess using ultrasound. For the ultrasound-guided infiltration method, a sterile linear probe with a 20 G guide was used to visualize the joint suprapatellar recess and avoid intrasynovial infiltration. The patient was positioned supine with the knee in full extension. From the lateral approach to the suprapatellar recess, HA was then injected into the knee joint, verifying intra-articular positioning in real-time via ultrasound imaging (direct visualization of viscous fluid or air bubbles).
  Patients did not receive anti-inflammatory or pain-relieving drugs in the week before the first injection . Patients were evaluated at four time points: at baseline and after 28, 42, 84, and 168 days after the intervention. At each evaluation, clinical data relating to the status of the disea

SUMMARY:
The prevalence of knee osteoarthritis (OA) is rising worldwide, leading to disability and a reduced quality of life, particularly in elderly patients. While there are several treatment options, there is little consensus in the scientific community over which methods are most effective. Viscosupplementation with hyaluronic acid (HA) has been found to reduce pain in patients with knee OA over a period of up to 6 months, with little to no side effects. The aim of this prospective open-label, uncontrolled, observational, single-site study was to assess the efficacy and safety of a single hybrid HA injection over a period of 6 months in subpopulations of patients with low to severe symptomatic knee OA in everyday clinical practice.

Fifty patients who met the inclusion criteria participated in the study. A single intra-articular ultrasound-guided injection of hybrid HA (Sinovial®) was administered. Patients submitted Visual Analog Scale (VAS) and Western Ontario and McMaster Universities Arthritis Index (WOMAC) questionnaires at 28-, 42-, 84-, and 168-days post-treatment.

ELIGIBILITY:
The inclusion criteria

1. medical indication for viscosupplementation therapy with hybrid HA 2 patients aged between 45 and 80 years 3.diagnosis of gonarthrosis 4. gonarthrosis symptoms for at least 6 months 5. patients who failed to respond to analgesics and/or regular NSAIDs, 6. grade 2 to 3 OA in the Kellgren-Lawrence grading scale 7. pain on walking measured by the Visual Analog Scale (VAS; 0-100 mm) of at least 40 mm on the targeted knee; 8. contralateral knee pain when walking with aVAS of less than 10 mm.

The exclusion criteria were:

1. inability to understand the aim of the study
2. inability to provide acceptable consent
3. pregnancy
4. serious psychiatric disorders
5. allergy or intolerance to hybrid HA
6. secondary gonarthrosis due to systematic and inflammatory disorders.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic OA of the knee KL II-III with unsucsessful conservative treatment with NSAIDS for 6 weeks. Age 45 -80 without axial deformation of the lower leg more than 10 deg.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 6 month
  Visual Analog Scale for the assessment of the pain during the study. Scale 0 ( no pain ) to 10 ( extreme pain )
The Western Ontario and McMaster Universities Arthritis Index | 6 months
  The Western Ontario and McMaster Universities Arthritis Index ( WOMAC ) is used to assess the function of the knee in osteoarthritis. Scale 0 ( the worst result ) -100 ( the best result )

CONTACTS AND LOCATIONS:
Locations (1):
- Sporto Clinic, Lodz, Poland

REFERENCES:
- [Derived] Domzalski ME, Marchewa K. The Efficacy and Safety of Single Injections of Hybrid HA in the Treatment of Symptomatic Knee Osteoarthritis: A Case Series. Rheumatol Ther. 2025 Aug;12(4):695-708. doi: 10.1007/s40744-025-00780-8. Epub 2025 Jul 2. PMID 40601162